CLINICAL TRIAL: NCT02461030
Title: An 8-Week Clinical Study to Evaluate the Efficacy of Two Oral Hygiene Regimens in the Reduction of Dentin Hypersensitivity After Non-surgical Periodontal Treatment: Randomized Clinical Trial
Brief Title: Efficacy of Two Oral Hygiene Regimens in the Reduction of Dentin Hypersensitivity After Periodontal Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Principal Investigator, Enilson Antonio Sallum, Professor, department of Periodontics, Piracicaba Dental School, State University of Campinas (UNICAMP), Piracicaba, São Paulo, Brazil, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 058/2013
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Dentin Sensitivity; Periodontal Diseases
Keywords: Dentin hypersensitivity; Periodontal disease; Arginine
MeSH Terms: conditions — Dentin Sensitivity; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CSPR + NS treatment (Experimental): In-office and at home Colgate sensitive pro-relief - CSPR
  Intervention: Non-surgical periodontal treatment (full-mouth debridement, scaling and root planing with ultrasonic/hand instruments) associated with In-office application of Colgate Sensitive Pro-Relief (CSPR) + tooth brushing with at home CSPR toothpaste during 8 weeks.
  Interventions: Drug: In-office and at home Colgate sensitive pro-relief - CSPR; Procedure: Non-surgical periodontal treatment
- Villevie® + NS treatment (Placebo Comparator): In-office Villevie® prophy paste + Colgate Toothpaste
  Treatment: In-office application of a Villevie® (fluoride-free) prophy paste + tooth brushing with a Colgate Cavity Protection Toothpaste during 8 weeks, after non-surgical periodontal treatment. (Full-mouth debridment/ Scaling and root planing with ultrasonic/hand instruments)
  Interventions: Drug: In-office Villevie® prophy paste + Colgate Toothpaste; Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Drug: In-office and at home Colgate sensitive pro-relief - CSPR — Prophylaxis with rubber cup using In-office Colgate sensitive pro-relief (CSPR), after non-surgical periodontal therapy, and tooth brushing with at home CSPR toothpaste.
  Other Names: CSPR
  Arms: CSPR + NS treatment
Drug: In-office Villevie® prophy paste + Colgate Toothpaste — Prophylaxis with rubber cup using In-office Villevie® (fluoride-free) prophy paste + Colgate Toothpaste, after non-surgical periodontal therapy.
  Other Names: Colgate Cavity Protection Toohtpaste
  Arms: Villevie® + NS treatment
Procedure: Non-surgical periodontal treatment — Full-mouth debridment, scaling and root planing with ultrasonic/hand instruments

SUMMARY:
This study aim is to determine the efficacy of two Oral Hygiene Regimens in the reduction of dentin hypersensitivity on subjects undergoing non-surgical periodontal treatment, over a period of 8 weeks.

DETAILED DESCRIPTION:
This study aim was to determine the efficacy of two Oral Hygiene Regimens in the reduction of dentin hypersensitivity on subjects undergoing non-surgical periodontal treatment, over a period of 8 weeks. The study was conducted in Piracicaba Dental School, Piracicaba, São Paulo, Brazil, using a double-blind/two treatment design. Sixty subjects (30 per group) that meet the inclusion and exclusion criteria were assigned to the groups: Test group (Non-surgical periodontal treatment + In-office application of Colgate Sensitive Pro-Relief - CSPR + tooth brushing with at home CSPR toothpaste) and Control group (Non-surgical periodontal treatment + In-office application of a fluoride-free prophy paste + tooth brushing with a Colgate Cavity Protection Toothpaste). Air blast sensitivity assessments were used to compare the efficacy of the two approaches using both the Schiff scale. The sensitivity parameters were measured at baseline, 1, 4 and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, between 30-75 years of age;
2. Availability for the duration of the study;
3. Individuals diagnosed with moderate chronic periodontal disease (4-5 mm loss of clinical attachment, according to AAP), and indication for non-surgical periodontal therapy;
4. Diagnosis, by air blast, of at least two (2) hypersensitive teeth with a score of 2 or 3 on the Schiff Cold Air Sensitivity Scale;
5. Subjects in good general health and no allergies to products that are being tested.

Exclusion Criteria:

1. Oral pathology, chronic disease, or a history of allergy to testing products;
2. Qualifying sensitive teeth with extensive/defective restorations, pulpitis, caries, cracked enamel, or these teeth used as abutments for removable partial dentures;
3. Subject using anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory medication or daily analgesics within one month prior to the start of the study or scheduled to start such intake during the course of the study;
4. Subject regularly using desensitizing toothpaste;
5. Current smokers;
6. Subject pregnant or breast feeding;
7. Allergies to oral care products, personal care consumer products, or their ingredients.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Dentin hypersensitivity reduction | Baseline, 8 weeks
  Air blast sensitivity assessments using Schiff scale at baseline and up to 8 weeks after non-surgical periodontal treatment.

SECONDARY OUTCOMES:
Probing depth reduction | Baseline, 8 weeks
  Full-mouth probing, at baseline and up to 8 weeks after non-surgical periodontal treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Enilson A Sallum, PhD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Piracicaba Dental School, State University of Campinas, Piracicaba, São Paulo, Brazil